CLINICAL TRIAL: NCT00585884
Title: Core Gel Study of the Safety and Effectiveness of Mentor Round Low Bleed Gel-filled Mammary Prostheses in Patients Who Are Undergoing Primary Breast Reconstruction or Revision
Brief Title: Following the Use of Gel Prosethetics in Breast Reconstruction
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Mentor Worldwide, LLC (Industry)
Responsible Party: Principal Investigator, Gregory R. Evans, Professor, University of California, Irvine
Other Study IDs: 20001383
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
Keywords: Reconstruction, Silicone prostheses
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Following placement of silicone breast prosthetics for reconstruction

DETAILED DESCRIPTION:
Patients undergoing breast reconstruction will be followed for outcomes after placement of silicone prostheses

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing breast surgery

Exclusion Criteria:

* Collagen vascular disease, Scleroderma

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women over 18 undergoing breast reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2001-02-01 (Actual); Primary Completion 2013-09-23 (Actual); Study Completion 2013-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Lewis, Study Chair — Mentor Worldwide, LLC
Locations (1):
- The University of California Irvine, Orange, California, United States